CLINICAL TRIAL: NCT02756468
Title: Procalcitonin Reveals Early Dehiscence in Pancreatic Surgery: the PREDIPS Study
Acronym: PREDIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Valentina Giaccaglia, MD, University of Roma La Sapienza
Other Study IDs: PREDIPS
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; procalcitonin
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pts operated for pancreatic cancer: all pts operated of pancreatic resection for cancer in the involved units
  Interventions: Other: pts operated for pancreatic cancer

INTERVENTIONS:
Other: pts operated for pancreatic cancer — measuring CRP and PCT in 3rd and 5th POD after pancreatic cancer resection

SUMMARY:
Background. Pancreatic cancer surgery is associated with very high risk of postoperative morbidity and mortality. Anastomotic leak (AL) is one of the worst complications associated with relevant short and long-term sequelae. Procalcitonin (PCT) is a biomarker used to monitor bacterial infections and guide antibiotic therapy and has been shown to have better predictive value of AL after colorectal surgery than C-reactive protein (CRP) and white blood cell count (WBC).

Purpose. The investigators designed a monocentric pilot study to test if PCT might be a sensitive and reliable marker of AL after pancreatic surgery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing all different kinds of pancreatic surgery
* in elective setting
* for cancer
* with a pancreatic anastomosis performed.

Exclusion Criteria:

* age < 18 years
* pregnant women
* patients undergoing pancreatic surgery for benign disease, other kinds of pancreatic surgery without an anastomosis being performed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all pts undergoing pacreatic resections for cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of PCT and CRP for anastomotic leak (AL) after pancreatic surgery | 2 yrs
  Sensitivity: % of patients corrected identified by the biomarkers having AL; PCT: procalcitonin, CRP: C-reactive protein, AL: anastomic leak
Specificity of PCT and CRP for anastomotic leak (AL) after pancreatic surgery | 2 yrs
  Specificity: % of pts corrected identified by the biomarkers not having AL; PCT: procalcitonin, CRP: C-reactive protein, AL: anastomic leak

SECONDARY OUTCOMES:
PCT and CRP cuts-off in 3rd POD with a good NPV for AL | 2 yrs
  PCT: procalcitonin, CRP: C-reactive protein, NPV: negative predictive value
PCT and CRP cuts-off in 5th POD with a good NPV for AL | 2 yrs
  PCT: procalcitonin, CRP: C-reactive protein, NPV: negative predictive value

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Andrea University Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No